CLINICAL TRIAL: NCT02664168
Title: A Prospective, Randomized, Comparative Study to Assess the Prevention of Surgical Site Infection (SSI's) in Revision Total Joint Arthroplasty Patients Treated With Single-Use Negative Pressure Wound Therapy (PICO™) or Standard Care Dressings (AQUACEL® Ag SURGICAL Dressing)
Brief Title: A Comparative Study to Assess the Prevention of Surgical Site Infection (SSI's) in Revision Total Joint Arthroplasty Patients Treated With Single-Use Negative Pressure Wound Therapy (PICO™) or Standard Care Dressings (AQUACEL® Ag SURGICAL Dressing)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Prevention
Other Study IDs: 2016Jpar01
Record Dates: First submitted 2016-01-22; First posted 2016-01-26 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Surgical Wound Infection
MeSH Terms: conditions — Surgical Wound Infection

ARMS (2):
- Aquacel Ag Surgical Dressing (Active Comparator)
  Interventions: Device: Aquacel Ag Surgical Dressing
- Single-Use Negative Pressure Wound Therapy (PICO) (Active Comparator)
  Interventions: Device: Single-Use Negative Pressure Wound Therapy (PICO)

INTERVENTIONS:
Device: Aquacel Ag Surgical Dressing
  Arms: Aquacel Ag Surgical Dressing
Device: Single-Use Negative Pressure Wound Therapy (PICO)
  Arms: Single-Use Negative Pressure Wound Therapy (PICO)

SUMMARY:
The aim of this study is to assess the prevention of incision healing complications in patients undergoing revision TKA and THA treated with either Single-Use NPWT (PICO) compared to standard of care dressings (AQUACEL Ag Surgical Dressing). All patients undergoing a revision TKA and THA who consent to taking part in the study, and meet the eligibility criteria will be included onto the study. Patients will be followed up for a period of up to 3 months to determine if there are any latent incision healing complications

ELIGIBILITY:
Inclusion Criteria:

1. Patient ≥18 years old
2. Male or non-pregnant, non-lactating, postmenopausal or surgically sterilized females
3. Subjects undergoing revision total knee arthroplasty or revision total hip arthroplasty
4. Subjects provide informed consent, which will consist of reading, signing, and dating the informed consent document after the Investigator, sub-Investigator or other designated study staff member has explained the study procedures, risks, and contact information
5. Subjects deemed able to understand and comply with study visit schedule and procedures

Exclusion Criteria:

1. Wounds that require daily inspection
2. Active bleeding within the surgical site
3. Pregnant, lactating females, or females of childbearing potential not willing to practice an effective method of contraception
4. Subjects on warfarin therapy. Resulting in increased exudate and prolonging hospital stay following surgery to achieve therapeutic INR levels
5. Skin integrity issues that preclude the use of Negative Pressure Wound Therapy (NPWT)
6. Subjects undergoing primary total joint procedures
7. Subjects with a known history of poor compliance with medical treatment
8. Subjects who have participated in this trial previously and who were withdrawn 9 . Subjects with known allergies to product components (silicone adhesives and polyurethane films (direct contact with wound), acrylic adhesives (direct contact with skin), polyethylene fabrics and super-absorbent powders (polyacrylates) (within the dressing)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2016-01; Primary Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of Surgical Site Infection | 90 days post-op

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Institute, Philadelphia, Pennsylvania, United States